CLINICAL TRIAL: NCT06596577
Title: Improving the Delivery and Equity of Inpatient Palliative Care: a Hybrid Type I Pragmatic Cluster Trial
Brief Title: Nudging Effective and Equitable Delivery of Specialty Palliative Care
Acronym: NEEDS-PC
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Katherine Courtright, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 856359; 1R01AG082874-01A1 (NIH)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Serious Illness; Palliative
Keywords: Palliative Care; Pragmatic Trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Palliative care needs information provision (Active Comparator): Clinicians will receive an EHR alert providing information about a patient's serious illness diagnosis(-es) and unmet palliative care needs
  Interventions: Behavioral: Palliative care needs information
- Palliative care needs information provision + default consult order (Active Comparator): The palliative care needs information provision intervention will be supplemented with a default palliative care consult order such that clinicians will receive an EHR alert providing information about a patient's serious illness diagnosis(-es) and unmet palliative care needs, and offered the choice to cancel the default consult order.
  Interventions: Behavioral: Default consult order
- Control/Usual Care (No Intervention): During the control phase, patients meeting eligibility criteria will be enrolled for study data collection but there will be no attempt to influence delivery of care. All hospitals will contribute a minimum of 9 weeks of outcomes data prior to adopting the intervention. The total duration of the control phase will differ for each hospital dependent on their randomly assigned time to adopt Intervention 1 in this stepped-wedge trial design.

INTERVENTIONS:
Behavioral: Palliative care needs information — clinician-directed EHR alert providing information about serious illness diagnosis(-es) and unmet palliative care needs
  Other Names: PC needs information
  Arms: Palliative care needs information provision
Behavioral: Default consult order — clinician-directed EHR alert providing information about serious illness diagnosis(-es) and unmet palliative care needs + a choice to cancel the default palliative care consult order
  Arms: Palliative care needs information provision + default consult order

SUMMARY:
This stepped-wedge, cluster randomized pragmatic trial among 9 MedStar hospitals for patients with serious illness and unmet palliative care (PC) needs will test two interventions embedded within the electronic health record (EHR): (1) a PC needs triggered alert to opt-in to PC consults nudging hospital clinicians to order specialty PC consults for eligible inpatients, and (2) a palliative care needs triggered alert with an opt-out to palliative care consults. The trial will compare the interventions effects to usual care, focusing on completed PC consults during the hospital encounter and other secondary outcomes. The trial also includes an embedded mixed methods study to explore factors influencing the effectiveness and equity of intervention implementation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older; AND
2. Admitted to inpatient status at 1 of the 9 participating hospitals
3. Meets validated score threshold of 8 from the MedStar unmet PC needs patient identification algorithm, utilizing empirically-derived weights for each PC need domain within the algorithm.

Exclusion Criteria:

1. Primary inpatient service: hospice, rehabilitation, psychiatry, obstetrics, neonatal
2. Signed hospital discharge order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18000 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Inpatient palliative care consultation | from enrollment up to 26 weeks
  Binary: at least 1 inpatient visit from a PC specialist during the hospital encounter

SECONDARY OUTCOMES:
Hospice enrollment | enrollment through 6 months
  Binary: hospice enrollment (any level of service)
Hospice duration | enrollment through 6 months
  Continuous: total days enrolled in hospice (any level of service)
Community palliative care referral | enrollment through 6 months
  Binary: order for community (home or outpatient clinic) palliative care consultation
Hospital all-cause mortality | enrollment to 1 day after hospital discharge
  Binary: (primary definition) death in the hospital; (secondary/sensitivity definition) death in the hospital or within 1 calendar day of discharge day.
30-day hospital readmission | hospital discharge through 30 days
  Binary: date of admission to an acute care hospital is within 30 days of hospital discharge
Number of readmissions | enrollment through 6 months
  Count: number of acute care hospital admissions
Hospital-free days | Enrollment through 6 months
  Count: days from enrollment spent alive and not in an acute care hospital through 6 months or death
Change in code status | from enrollment up to 26 weeks
  Binary; any change in code status order at enrollment and code status order at hospital discharge
Time to palliative care consult | from enrollment up to 26 weeks
  Continuous (hours): enrollment to documentation timestamp of first inpatient palliative care consult
Discharge to hospice | from enrollment up to 26 weeks
  Binary: (primary definition) hospital discharge disposition to hospice (any location or level of service); (secondary/sensitivity analysis definition) hospital discharge disposition to hospice or comfort-focused care orders in-hospital
Hospital length of stay | from enrollment up to 26 weeks
  Continuous: enrollment time to hospital discharge order timestamp.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Courtright, MD, MS, Principal Investigator — University of Pennsylvania; Michael Harhay, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (9):
- United States (9):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Health Center, Washington D.C., District of Columbia
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Harbor Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - MedStar St. Mary's Hospital, Leonardtown, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to researchers upon request and approval by the study investigators of a valid research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data generated from this project will be made available no later than 1 year after publication of the primary trial manuscript.
Access Criteria: Proposals for data use will be reviewed by Principal Investigator and independent review boards (such as Institutional Review Board, Data Safety and Monitoring Board, and a Stakeholder Advisory Committee). Approved data requestors will need to sign data use agreements to access and use de-identified data.